CLINICAL TRIAL: NCT07063745
Title: A Randomized Phase 2/3 Study of BMS-986504 in Combination With Pembrolizumab and Chemotherapy Versus Placebo Plus Pembrolizumab and Chemotherapy in First-line Metastatic Non-small Cell Lung Cancer Participants With Homozygous MTAP Deletion
Brief Title: A Study to Compare the Combination of BMS-986504 With Pembrolizumab and Chemotherapy Versus Placebo Plus Pembrolizumab and Chemotherapy in First-line Metastatic Non-small Cell Lung Cancer Participants With Homozygous MTAP Deletion
Acronym: MountainTAP-29
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA240-0029; 2025-521511-40 (Other: EU CT Number); U1111-1319-8383 (Other: UTN); CA2400029 (Other: Bristol-Myers Squibb Protocol ID)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Non-small Cell Lung Cancer With MTAP Deletion
Keywords: PRMT5; Lung cancer; NSCLC; MTAP; CDKN2A; MRTX1719; First-line
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Phase 2 portion of this study will be blinded to sites, participants, investigators, and certain site-facing members of the Sponsor.
  The Phase 3 portion of this study will be blinded to participants, investigators, and the Sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A: BMS-986504 + Pembrolizumab + Chemotherapy (Active Comparator)
  Interventions: Drug: BMS-986504; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm B: BMS-986504 + Pembrolizumab + Chemotherapy (Active Comparator)
  Interventions: Drug: BMS-986504; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm C: Placebo + Pembrolizumab + Chemotherapy (Placebo Comparator)
  Interventions: Drug: Pembrolizumab; Other: Placebo; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm D: Placebo + Pembrolizumab + Chemotherapy (Placebo Comparator)
  Interventions: Drug: Pembrolizumab; Other: Placebo; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm E: BMS-986504 + Pembrolizumab + Chemotherapy (Active Comparator)
  Interventions: Drug: BMS-986504; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm F: Placebo + Pembrolizumab + Chemotherapy (Placebo Comparator)
  Interventions: Drug: Pembrolizumab; Other: Placebo; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: BMS-986504 — Specified dose on specified days
  Arms: Arm A: BMS-986504 + Pembrolizumab + Chemotherapy; Arm B: BMS-986504 + Pembrolizumab + Chemotherapy; Arm E: BMS-986504 + Pembrolizumab + Chemotherapy
Drug: Pembrolizumab — Specified dose on specified days
Other: Placebo — Specified dose on specified days
  Arms: Arm C: Placebo + Pembrolizumab + Chemotherapy; Arm D: Placebo + Pembrolizumab + Chemotherapy; Arm F: Placebo + Pembrolizumab + Chemotherapy
Drug: Cisplatin — Specified dose on specified days
Drug: Carboplatin — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Paclitaxel — Specified dose on specified days
Drug: Nab-paclitaxel — Specified dose on specified days

SUMMARY:
The purpose of this study is to compare the clinical benefit of the combination of BMS-986504 (a selective MTA-cooperative inhibitor of PRMT5) plus pembrolizumab and chemotherapy versus placebo plus pembrolizumab and chemotherapy in first-line metastatic non-small cell lung cancer participants with homozygous MTAP deletion

ELIGIBILITY:
Inclusion Criteria

* Participants must have Metastatic (Stage IV or recurrent) non-small cell lung cancer (NSCLC) (as defined by the American Joint Committee on Cancer, Ninth Edition) with no prior systemic anti-cancer therapy for metastatic disease.
* Participants must have histologically confirmed diagnosis of NSCLC and homozygous methylthioadenosine phosphorylase (MTAP) deletion or MTAP loss.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Participants must have at least 1 measurable lesion as per RECIST v1.1.

Exclusion Criteria

* Nonsquamous participants must not have documented targetable oncogenic mutation or actionable genetic alterations (AGAs) for which there is a standard of care (SoC) available as first-line (1L) therapy.
* Participants must not have symptomatic brain metastases or spinal cord compression.
* Participants must not have any prior systemic therapy (chemotherapy, immunotherapy, targeted therapy, or biological therapy) for metastatic non-small cell lung cancer (mNSCLC). Note: One cycle of SoC treatment prior to randomization will be allowed for participants who require immediate treatment if clinically indicated.
* Participants must not have any known or suspected impairment of gastrointestinal function that may prohibit the ability to absorb or swallow an oral medication without chewing or crushing.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2031-08-12 (Estimated); Study Completion 2031-08-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
Overall Survival (OS) | Up to 5 years
  Phase 3

SECONDARY OUTCOMES:
Objective response (OR) (confirmed complete response (CR) or partial response (PR)) | Up to 2 years
  Phase 2
Disease control (best overall response (BOR) of confirmed CR, confirmed PR, or stable disease (SD)) | Up to 2 years
  Phase 2
Time to objective response (TTOR) (CR or PR) | Up to 2 years
  Phase 2
Duration of response (DOR) (CR or PR) | Up to 2 years
  Phase 2
OR (confirmed CR or PR) | Up to 5 years
  Phase 3
Disease control (BOR of confirmed CR, confirmed PR, or SD) | Up to 5 years
  Phase 3
DOR (CR or PR) | Up to 5 years
  Phase 3
PFS | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (259):
- United States (34):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Local Institution - 0388, Phoenix, Arizona
  - Local Institution - 0120, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Local Institution - 0407, Los Angeles, California
  - Local Institution - 0444, Los Angeles, California
  - Local Institution - 0152, Fort Lauderdale, Florida
  - Local Institution - 0389, Jacksonville, Florida
  - Local Institution - 0430, St. Petersburg, Florida
  - St. Luke's Cancer Institute: Boise, Boise, Idaho
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Local Institution - 0127, Scarborough, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 0418, Ann Arbor, Michigan
  - Local Institution - 0405, Detroit, Michigan
  - Local Institution - 0420, Traverse City, Michigan
  - Local Institution - 0182, Rochester, Minnesota
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Local Institution - 0467, Lebanon, New Hampshire
  - Local Institution - 0179, Hawthorne, New York
  - Local Institution - 0128, Rochester, New York
  - Local Institution - 0163, Cleveland, Ohio
  - Local Institution - 0129, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente Interstate Medical Office Central, Portland, Oregon
  - Local Institution - 0433, Dallas, Texas
  - Local Institution - 0374, El Paso, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Local Institution - 0377, The Woodlands, Texas
  - Local Institution - 0354, Salt Lake City, Utah
  - Local Institution - 0131, Fairfax, Virginia
  - Local Institution - 0186, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Argentina (4):
  - Local Institution - 0465, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0463, Rosario, Santa Fe Province
  - Local Institution - 0447, Buenos Aires
  - Local Institution - 0446, Buenos Aires
- Australia (7):
  - Local Institution - 0432, Liverpool, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Local Institution - 0431, Hobart, Tasmania
  - Local Institution - 0367, Ballarat Central, Victoria
  - Local Institution - 0368, Garran
  - Local Institution - 0373, Woolloongabba
- Austria (3):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Landeskrankenhaus Rankweil, Rankweil
  - Local Institution - 0207, Vienna
- Belgium (6):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Local Institution - 0226, Hasselt, Limburg
  - Local Institution - 0225, Yvoir, Namur
  - AZ Delta vzw, Roeselare, West-Vlaanderen
  - UZ Brussel, Brussels
  - Local Institution - 0340, Liège
- Brazil (12):
  - Local Institution - 0088, Vitória, Espírito Santo
  - Local Institution - 0079, Natal, Rio Grande do Norte
  - Local Institution - 0346, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0085, Blumenau, Santa Catarina
  - Local Institution - 0081, Barretos, São Paulo
  - Local Institution - 0076, Bauru, São Paulo
  - Local Institution - 0094, Campinas, São Paulo
  - Local Institution - 0355, São Caetano do Sul, São Paulo
  - Local Institution - 0351, São José do Rio Preto, São Paulo
  - Local Institution - 0095, São Paulo, São Paulo
  - Local Institution - 0091, Rio de Janeiro
  - Local Institution - 0078, São Paulo
- Bulgaria (6):
  - Local Institution - 0315, Panagyurishte, Pazardzhik
  - Local Institution - 0459, Sofia, Sofia
  - Local Institution - 0309, Haskovo
  - Complex Oncology Center - Ruse EOOD, Rousse
  - Local Institution - 0460, Sofia
  - Local Institution - 0307, Stara Zagora
- China (39):
  - Local Institution - 0072, Hefei, Anhui
  - Local Institution - 0074, Beijing, Beijing Municipality
  - Local Institution - 0049, Beijing, Beijing Municipality
  - Local Institution - 0286, Beijing, Beijing Municipality
  - Local Institution - 0046, Fuzhou, Fujian
  - Local Institution - 0100, Xiamen, Fujian
  - Local Institution - 0099, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Local Institution - 0061, Guangzhou, Guangdong
  - Local Institution - 0281, Shenzhen, Guangdong
  - Guangxi Medical University Affiliated Cancer Hospital, Nanning, Guangxi
  - Local Institution - 0408, Guiyang, Guizhou
  - Local Institution - 0353, Shijiazhuang, Hebei
  - Local Institution - 0106, Harbin, Heilongjiang
  - Local Institution - 0107, Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center, Wuhan, Hubei
  - Local Institution - 0059, Wuhan, Hubei
  - Local Institution - 0387, Changsha, Hunan
  - Local Institution - 0050, Changsha, Hunan
  - Local Institution - 0352, Nanjing, Jiangsu
  - Local Institution - 0279, Nanjing, Jiangsu
  - Local Institution - 0110, Nanchang, Jiangxi
  - Local Institution - 0284, Shenyang, Liaoning
  - Local Institution - 0104, Shenyang, Liaoning
  - Local Institution - 0103, Shenyang, Liaoning
  - Local Institution - 0060, Xi'an, Shaanxi
  - Local Institution - 0051, Jinan, Shandong
  - Local Institution - 0066, Linyi, Shandong
  - Local Institution - 0068, Qingdao, Shandong
  - Local Institution - 0278, Shanghai, Shanghai Municipality
  - Local Institution - 0343, Shanghai, Shanghai Municipality
  - Local Institution - 0283, Taiyuan, Shanxi
  - Local Institution - 0102, Chengdu, Sichuan
  - Local Institution - 0109, Chengdu, Sichuan
  - Local Institution - 0280, Hangzhou, Zhejiang
  - Local Institution - 0069, Hangzhou, Zhejiang
  - Local Institution - 0054, Hangzhou, Zhejiang
  - Local Institution - 0386, Nanjing
  - Local Institution - 0047, Zhengzhou
- Colombia (3):
  - Local Institution - 0330, Medellín, Antioquia
  - Local Institution - 0305, Bogotá, Cundinamarca
  - Local Institution - 0306, Montería, Departamento de Córdoba
- Czechia (2):
  - Local Institution - 0251, Hradec Králové, Hradec Králové
  - Local Institution - 0250, Olomouc
- Local Institution - 0356, Copenhagen, Capital Region, Denmark
- France (17):
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Centre François Baclesse, Caen, Calvados
  - Local Institution - 0212, Dijon, Côte-d'Or
  - Chu Jean Minjoz, Besançon, Doubs
  - CHRU de Brest, Brest, Finistère
  - CHU de Toulouse - Hopital Larrey, Toulouse, Haute-Garonne
  - Local Institution - 0220, Montpellier, Hérault
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Local Institution - 0215, Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Chu Gabriel Montpied, Clermont-Ferrand, Puy-de-Dôme
  - Local Institution - 0214, Pierre-Bénite, Rhône
  - Local Institution - 0213, Créteil, Val-de-Marne
  - Local Institution - 0218, Paris
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
  - Local Institution - 0429, Paris, Île-de-France Region
- Germany (9):
  - Local Institution - 0461, Göppingen, Baden-Wurttemberg
  - Robert Bosch Krankenhaus GmbH, Stuttgart, Baden-Wurttemberg
  - Local Institution - 0462, Ulm, Baden-Wurttemberg
  - Local Institution - 0202, München, Bavaria
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg, Bavaria
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - LungenClinic Grosshansdorf, Großhansdorf
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinik Löwenstein, Löwenstein
- Greece (6):
  - Local Institution - 0008, Pátrai, Achaḯa
  - Local Institution - 0005, Athens, Attikí
  - Thoracic General Hospital of Athens "I Sotiria", Athens, Attikí
  - Local Institution - 0009, Athens, Attikí
  - Local Institution - 0006, Thessaloniki, Kentrikí Makedonía
  - University General Hospital of Larissa, Larissa, Thessalía
- Hong Kong (2):
  - Local Institution - 0285, Hksar
  - Local Institution - 0323, Shatin
- Hungary (4):
  - Local Institution - 0290, Gyula, Bekes County
  - Local Institution - 0291, Gyöngyös, Heves County
  - Local Institution - 0287, Farkasgyepű, Veszprém megye
  - Local Institution - 0288, Budapest
- India (7):
  - Local Institution - 0263, Bangalore, Karnataka
  - Local Institution - 0344, Bengaluru, Karnataka
  - Local Institution - 0345, Mumbai, Maharashtra
  - Local Institution - 0266, Mumbai, Maharashtra
  - Local Institution - 0267, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0265, Hyderabad, Telangana
  - Local Institution - 0264, Varanasi, Uttar Pradesh
- Israel (6):
  - Local Institution - 0010, Kfar Saba, Central District
  - Local Institution - 0011, Ramat Gan, Central District
  - Local Institution - 0017, Jerusalem, Jerusalem
  - Local Institution - 0013, Jerusalem, Jerusalem
  - Local Institution - 0016, Afula, Northern District
  - Local Institution - 0014, Haifa, Northern District
- Italy (8):
  - Local Institution - 0105, Napoli, Campania
  - Ospedale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Local Institution - 0037, Orbassano, Torino
  - Local Institution - 0044, Perugia, Umbria
  - Local Institution - 0098, Bologna
  - Local Institution - 0039, Milan
  - Ospedale San Raffaele, Milan
- Japan (20):
  - Local Institution - 0243, Nagoya, Aichi-ken
  - Local Institution - 0236, Kashiwa, Chiba
  - Local Institution - 0334, Otashi, Gunma
  - Local Institution - 0233, Sapporo, Hokkaido
  - Local Institution - 0336, Himeji, Hyōgo
  - Local Institution - 0247, Kobe, Hyōgo
  - Local Institution - 0335, Shiwa-gun Yahaba-cho, Iwate
  - Local Institution - 0257, Kawasaki, Kanagawa
  - Local Institution - 0238, Yokohama, Kanagawa
  - Local Institution - 0241, Nankoku, Kochi
  - Local Institution - 0237, Matsusaka, Mie-ken
  - Local Institution - 0232, Sendai, Miyagi
  - Local Institution - 0240, Hirakata, Osaka
  - Local Institution - 0245, Hidaka, Saitama
  - Local Institution - 0235, Shimotsuga, Tochigi
  - Local Institution - 0234, Bunkyo-ku, Tokyo
  - Local Institution - 0242, Ube, Yamaguchi
  - Local Institution - 0246, Fukuoka
  - Local Institution - 0244, Okayama
  - Local Institution - 0239, Osaka
- Malaysia (2):
  - Local Institution - 0413, Kuala Lumpur, Kuala Lumpur
  - Local Institution - 0390, Kuching, Sarawak
- Mexico (9):
  - Local Institution - 0296, Guadalajara, Jalisco
  - Local Institution - 0326, Guadalajara, Jalisco
  - Local Institution - 0293, Mexico City, Mexico City
  - Local Institution - 0294, Mexico City, Mexico City
  - Local Institution - 0298, Monterrey, Nuevo León
  - Local Institution - 0297, Oaxaca City, Oaxaca
  - Local Institution - 0328, Querétaro City, Querétaro
  - Local Institution - 0327, Chihuahua City
  - Local Institution - 0331, Puebla City
- Netherlands (3):
  - Local Institution - 0445, Veldhoven, North Brabant
  - Local Institution - 0230, Arnhem
  - University Medical Center Groningen, Groningen
- Local Institution - 0096, Drammen, Buskerud, Norway
- Poland (6):
  - Centrum Medyczne Pratia Poznań, Poznan, Greater Poland Voivodeship
  - Local Institution - 0259, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0261, Warsaw, Masovian Voivodeship
  - Local Institution - 0458, Wieliszew, Masovian Voivodeship
  - Local Institution - 0258, Prabuty, Pomeranian Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz
- Romania (9):
  - Institutul Oncologic Bucuresti "Prof. Dr. Alexandru Trestioreanu", Bucharest, București
  - Local Institution - 0019, Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Local Institution - 0027, Otopeni, Ilfov
  - Local Institution - 0020, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - S.C. Centrul de Oncologie Euroclinic S.R.L., Iași
  - Institutul Regional de Oncologie, Iași
  - Local Institution - 0030, Ploieşti
- South Korea (7):
  - Local Institution - 0272, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Local Institution - 0270, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0269, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (9):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0248, Hospitalet, Barcelona [Barcelona]
  - Local Institution - 0253, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0118, Madrid, Madrid, Comunidad de
  - Local Institution - 0254, Madrid, Madrid, Comunidad de
  - Local Institution - 0252, Majadahonda, Madrid, Comunidad de
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Local Institution - 0255, Valencia
- Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands Län [se-14], Sweden
- Taiwan (5):
  - Chi Mei Medical Center Liouying Branch, Tainan, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Thailand (2):
  - Local Institution - 0411, Bangkok
  - Local Institution - 0412, Bangkok
- Turkey (Türkiye) (7):
  - Local Institution - 0349, Izmir, Karsiyaka, İzmir
  - Local Institution - 0318, Adana
  - Local Institution - 0317, Adana
  - Local Institution - 0321, Ankara
  - Local Institution - 0350, Antalya
  - Local Institution - 0320, Bursa
  - Local Institution - 0319, Edirne
- United Kingdom (2):
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Sarah Cannon Research Institute UK, London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07063745.html